CLINICAL TRIAL: NCT04971759
Title: Addition of Dexmedetomidine to Levobupivacaine for Transversus Abdominis Plane Block in Elderly Patients Undergoing Inguinal Hernia Repair Surgery: Could it Make a Difference?
Brief Title: Dexmedetomidine to Levobupivacaine for Transversus Abdominis Plane Block in Elderly Patients Undergoing Inguinal Hernia Repair Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Mohammed AboelFadl, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17300618
Record Dates: First submitted 2021-07-06; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Dexmedetomidine; Fentanyl
MeSH Terms: interventions — Levobupivacaine; Dexmedetomidine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group L (Experimental): 30 Patients will receive Levobupivacaine 5%
  Interventions: Drug: Levobupivacaine
- LD group (Experimental): 30 patients will receive Levobupivacaine 5% + 1 µg/kg dexmedetomidine.
  Interventions: Drug: Dexmedetomidine Hydrochloride
- LF group (Experimental): 30 patients will receive Levobupivacaine 5% + 1µg/kg fentanyl
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Levobupivacaine — Levobupivacaine 5%
  Arms: Group L
Drug: Dexmedetomidine Hydrochloride — Levobupivacaine 5% + 1 µg/kg dexmedetomidine.
  Arms: LD group
Drug: Fentanyl — Levobupivacaine 5% + 1µg/kg fentanyl
  Arms: LF group

SUMMARY:
The perioperative management of pain following abdominal surgery can pose a challenge to anesthesia providers. Conventional practice has involved the use of opioids as well as neuraxial analgesic techniques. Unfortunately, these therapies are not without potential risks and side effects. These include nausea, vomiting, pruritus, urinary retention, constipation, respiratory depression, and sedation.

DETAILED DESCRIPTION:
As a result, the goal to reduce perioperative pain has taken on a multimodal approach.

Multimodal or "balanced" analgesia uses a combination of opioid and nonopioid analgesics to improve pain control and minimize opioid-related side effects. These include the use of nonsteroidal anti-inflammatory drugs, local anesthetics, peripheral nerve blocks, gabapentinoids, and alpha2 adrenergic agonists. Any combination of these therapies can help reduce the surgical stress response and improve patient outcomes such as pain control, patient satisfaction, time to discharge, and return to daily activities.

One method used in this multimodal approach is the transversus abdominis plane block. As first described by Rafi in 2001, this block provides analgesia to the anterolateral abdominal wall. In 2007, further studied this technique in patients undergoing large-bowel resection. He discovered a reduction in postoperative pain and morphine consumption in the first 24 hours postoperatively, resulting in fewer opioid-mediated side effects. In this same year, Hebbard described the use of ultrasound guidance to provide real-time imaging of the muscle layers and needle placement to improve TAP block accuracy. In 2008, Hebbard. described the subcostal approach of TAP blocks, to target the nerves of the upper abdomen. Transversus abdominis plane blocks continue to be studied and developed as an effective method for providing analgesia for numerous types of abdominal surgeries.

ELIGIBILITY:
Inclusion Criteria:

* ASA status I, II, and III patients,
* aged 60-75 y,
* both male and female,
* undergoing inguinal hernia repair surgery.

Exclusion Criteria:

* morbid obesity (BMI > 40),
* spine metastatic tumor, allergy to an amide LA, or magnesium sulfate,
* heart block, renal, or liver dysfunction, substance abuse disorder, chronic opioid use, or electrolyte disturbance, administration of any sedative, preexisting mental illness, psychological or emotional problems.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
first analgesic request | 24 hours postoperative
  time for the first analgesia rescue call.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut governorate, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Milone M, Di Minno MN, Musella M, Maietta P, Salvatore G, Iacovazzo C, Milone F. Outpatient inguinal hernia repair under local anaesthesia: feasibility and efficacy of ultrasound-guided transversus abdominis plane block. Hernia. 2013 Dec;17(6):749-55. doi: 10.1007/s10029-012-1022-2. Epub 2012 Nov 16. PMID 23160979
- [Result] Favuzza J, Brady K, Delaney CP. Transversus abdominis plane blocks and enhanced recovery pathways: making the 23-h hospital stay a realistic goal after laparoscopic colorectal surgery. Surg Endosc. 2013 Jul;27(7):2481-6. doi: 10.1007/s00464-012-2761-y. Epub 2013 Jan 26. PMID 23355160
- [Result] Walter CJ, Maxwell-Armstrong C, Pinkney TD, Conaghan PJ, Bedforth N, Gornall CB, Acheson AG. A randomised controlled trial of the efficacy of ultrasound-guided transversus abdominis plane (TAP) block in laparoscopic colorectal surgery. Surg Endosc. 2013 Jul;27(7):2366-72. doi: 10.1007/s00464-013-2791-0. Epub 2013 Feb 7. PMID 23389068